CLINICAL TRIAL: NCT05769569
Title: Safety and Efficacy of Broadly Neutralizing Antibodies Followed by Innate Immune Stimulation and Therapeutic Vaccination for the Induction of HIV Remission
Brief Title: Safety and Efficacy of Neutralizing Antibodies and Vaccination for Induction of HIV Remission
Acronym: RV582
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol was changed during development
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: US Military HIV Research Program (Network); Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RV 582
Record Dates: First submitted 2023-02-15; First posted 2023-03-15 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: HIV-1-infection
Keywords: human immunodeficiency virus-1; PLWH; AHI; ART; HIV-1; antiretroviral therapy; acute HIV-1 infection
MeSH Terms: interventions — ALT-803; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Intervention Model Description: This is a phase I, randomized, open-label trial to investigate the safety of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination, and the impact on time to sustained viral rebound of ≥1000 copies/mL for 4 consecutive weeks during ATI in PLWH who initiated ART during AHI. The study will involve 35 adults who initiated ART during Fiebig I-V acute HIV infection, with plasma HIV RNA <50 copies/mL for ≥48 weeks, CD4 T-cell counts ≥450 cells/mm3, viruses susceptible to both VRC07-523LS and PGDM1400LS and the absence of known protective HLA allele.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antiretroviral therapy + Investigational Products (Experimental): Active Group (ART with the addition of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV, A244d11 gp120 and ALFQ vaccination)
  Interventions: Biological: VRC07-523LS; Biological: PGDM1400LS; Biological: N-803; Biological: Ad26.Mos4.HIV; Biological: MVA-BN-HIV; Biological: A244d11 gp120; Biological: ALFQ; Combination Product: Antiretroviral Therapy (ART)
- Antiretroviral therapy only (Active Comparator): Control Group (continue only with ART without further interventions)
  Interventions: Combination Product: Antiretroviral Therapy (ART)

INTERVENTIONS:
Biological: VRC07-523LS — VRC07-523LS is a recombinant human immunoglobulin G1 (IgG1) broadly neutralizing monoclonal antibody (bNAb) directed against the HIV-1 CD4 binding site. Intravenous infusion of 10 mg/kg VRC07-523LS will be administered on Week 0.
  Other Names: VRC-HIVMAB075-00-AB
  Arms: Antiretroviral therapy + Investigational Products
Biological: PGDM1400LS — PGDM1400LS is a recombinant human IgG1 bNAb targeted against the HIV-1 V2 apex epitope region. Intravenous infusion of 20 mg/kg PGDM1400LS will be administered on Week 0.
  Arms: Antiretroviral therapy + Investigational Products
Biological: N-803 — N-803 is a recombinant human superagonist interleukin-15 (IL-15) complex. N-803 at 6 ug/kg will be administered via subcutaneous injection to the trunk on Weeks 1, 4, 7, 39, 42 and 45.
  Arms: Antiretroviral therapy + Investigational Products
Biological: Ad26.Mos4.HIV — Ad26.Mos4.HIV is a tetravalent vaccine comprising Ad26.Mos1.Env, Ad26.Mos2S.Env, Ad26.Mos1.Gag-Pol, and Ad26.Mos2.Gag-Pol. Ad26.Mos4.HIV at 5x1010 viral particles (per 0.5 mL dose) will be administered through intramuscular injection in the quadriceps muscle at Week 11.
  Arms: Antiretroviral therapy + Investigational Products
Biological: MVA-BN-HIV — MVA-BN-HIV is a single vector recombinant Modified Vaccinia Ankara - Bavarian Nordic (MVA-BN®) expressing Mos1.Env, Mos2S.Env, Mos1.Gag-Pol, and Mos2.Gag-Pol. MVA-BN-HIV at 2x108 infectious unit (per 0.5mL dose) will be administered through intramuscular injection in the quadriceps muscle at Week 35.
  Arms: Antiretroviral therapy + Investigational Products
Biological: A244d11 gp120 — A244d11 gp120, consists of the gp120 envelope glycoprotein HIV-1 subtype CRF_01AE A244 derived from the CM244 CRF_01AE strain, with an 11 amino N-terminal deletion. It is a modification of the A244 rgp120 immunogen from the AIDSVAX®B/E vaccine. A244d11 gp120 at 300 ug will be administered as an intramuscular injection in the quadriceps muscle at week 11 and week 35.
  Arms: Antiretroviral therapy + Investigational Products
Biological: ALFQ — ALFQ (Army Liposome Formulation, ALF) is a liposomal adjuvant containing a synthetic monophosphoryl lipid A (MPLA, 3D-PHAD®) with the addition of QS-21. ALFQ at 200 ug will be administered as an intramuscular injection in the quadriceps muscle at week 11 and week 35.
  Arms: Antiretroviral therapy + Investigational Products
Combination Product: Antiretroviral Therapy (ART) — This study will enroll PLWH aged 18-50 years who initiated ART during Fiebig I-V AHI and are virologically suppressed (HIV RNA <50 copies/ml for ≥48 weeks) on uninterrupted ART, who meet study inclusion criteria in Bangkok, Thailand.

SUMMARY:
This is a phase I, randomized, open-label trial to investigate the safety of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-Bavarian Nordic (BN)-HIV and A244d11gp120/ALFQ vaccination, and the impact on time to sustained viral rebound of ≥1000 copies/mL for 4 consecutive weeks during analytic treatment interruption (ATI) in people living with human immunodeficiency virus-1 (HIV-1, PLWH) who initiated antiretroviral therapy (ART) during acute HIV-1 infection (AHI).

DETAILED DESCRIPTION:
This is a phase 1 study. The study duration is approximately 134 weeks. The primary objectives are:

1. To evaluate the safety of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination in PLWH who initiated ART during AHI.
2. To evaluate the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on time to sustained viral rebound to ≥1000 copies/mL for 4 consecutive weeks AND has not declined by >0.2 log10 from the previous measurement during ATI.

ELIGIBILITY:
Step 1 Inclusion Criteria

Participants are eligible to be included in the protocol Step 1 only if all of the following criteria are met:

1. Thai National
2. Age ≥18 and ≤50 years of age
3. Can read and write Thai or English
4. Able and willing to provide written informed consent
5. Participant of the RV254 study
6. Confirmed HIV-1 infection (nucleic acid testing [NAT] and/or HIV serology positive with confirmatory quantitative HIV viral load) and started ART during acute infection (Fiebig stage I-V)
7. Uninterrupted treatment with ART (no interruption of ART for ≥7 consecutive days or longer) since ART initiation, for ≥ 48 weeks.
8. Currently on integrase inhibitor-based ART regimen (excluding long-acting injectable regimens) and no recent (≤8 weeks prior to screening) changes to ART regimen.

   a. There must be at least one documented plasma HIV RNA <50 cps/mL after the last ART change prior to screening
9. Must be medically stable as confirmed by medical history, physical examination, vital signs, and clinical laboratory tests performed at screening, and as per the Investigator's discretion.

   a. If the results of the screening laboratory panel (except those listed specifically in inclusion criterion) are outside the normal reference ranges, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study after discussion with the Sponsor's Representative.
10. The following laboratory values at screening:

    1. Absolute neutrophil count (ANC) ˃1,000/mm3
    2. Hemoglobin >11.5 g/dL
    3. Platelet count ˃150,000/mm3
    4. Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 using the re-expressed MDRD equation with Thai racial factor or the CKD-EPI Cystatin C equation.
    5. Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and alkaline phosphatase (AP) ≤1 x ULN
    6. Total bilirubin ≤1 x ULN
    7. Troponin <1 x ULN
11. HIV RNA <50 copies/ml for ≥48 weeks at screening.

    1. No history of virologic failure. Virologic failure is defined as having two consecutive HIV-1 RNA >1000 copies/mL at any time after achieving HIV-1 RNA <50 copies/mL.
    2. A single viral load measurement ≥50 but <1000 copies/mL, at any time from achieving HIV-1 RNA <50 copies/mL to > 48 weeks from screening, is allowed provided that it is bracketed by viral loads <50 copies/mL.
    3. A single viral load measurements ≥50 but <200 copies/mL, within 48 weeks of screening is allowed provided that each is bracketed by viral loads <50 copies/mL prior to screening.
12. CD4 T-cell count ≥450 cells/mm3 at screening.
13. Sensitivity test demonstrating the lack of detection of resistant viruses to VRC07-523LS and PGDM1400LS
14. For persons of childbearing potential, negative pregnancy test at the screening visit.
15. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy. One contraceptive method must be from the list of highly effective methods listed in section 7.5.3 of the protocol. The second method of contraception must be from the barrier methods also listed in section 7.5.3.Contraception must be used from the time of screening to the end of study .
16. Participants engaging in sexual activity that could lead to pregnancy in the partner and who are of reproductive potential must agree to use a condom to avoid pregnancy in a spouse or partner of childbearing potential and to avoid transmitting HIV to an uninfected partner. A condom must be used from the time of screening until the end of the study.
17. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using pre-exposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
18. Passes Test of Understanding (Section 8.4)
19. Willing to interrupt and restart ART according to study schedule
20. Willing to participate and adhere to the prohibitions and restrictions specified in this protocol for the duration of the study visits and follow up.

Step 1 Exclusion Criteria

Participants who meet any of the following criteria will be excluded from the study:

1. Weight <50 kg or > 115 kg
2. Presence of HLA allele associated with viral control including HLA B*57:01 or HLA B*58:01 (based on archived data from RV254)
3. Anyone with contraindication to intramuscular injections, placement of intravenous lines, and blood draws
4. Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to entry.
5. Any clinically significant acute or chronic medical condition, that in the opinion of the investigator would preclude participation including cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological disorders, that in the opinion of the investigator would preclude participation (e.g., history of seizure disorders, cardiovascular disease, bleeding/clotting disorder, autoimmune disease, malignancy, poorly controlled asthma, active tuberculosis or other systemic infections, etc.)

   1. Participants with acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) including untreated syphilis, gonorrhea or chlamydia infection or temperature ≥38.0ºC within 24 hours prior to the first dose of IP will not enter baseline. Participant will be referred for treatment, and participant is eligible for repeat screening and potential study entry once treatment is successfully completed
   2. Major surgery (per the Investigator's judgment) within 12 weeks before screening or plan to have major surgery during the time of study participation

      • surgical procedures to be conducted under local or loco-regional anesthesia and not judged as major by the Investigator may participate.
   3. Current or history of an HIV-associated malignancy (including Kaposi's sarcoma), and any type of lymphoma, or virus-associated cancers
   4. Current or history of non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the 36 months prior to screening

      • Minor surgical removal of localized skin cancers (squamous cell carcinoma, basal cell carcinoma) or carcinoma in situ of the cervix is not exclusionary
   5. Current or history of clinical atherosclerotic cardiovascular disease, as defined by 2013 American College of Cardiology (ACC)/American Heart Association (AHA) guidelines, including a previous diagnosis of any of the following: acute myocardial infarction, acute coronary syndromes, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack (TIA), peripheral arterial disease presumed to be of atherosclerotic origin
   6. Current or history of myocarditis, pericarditis, cardiomyopathy, congestive heart failure with permanent sequelae, clinically significant arrhythmia (including any arrhythmia requiring medication, treatment, or clinical follow-up)
   7. Current or history of advanced liver disease (non-alcoholic fatty liver disease, steatohepatitis, or alcoholic liver disease) with known or suspected cirrhosis or fibrosis score ≥F2.
   8. Current or history of TTS, or heparin-induced thrombocytopenia and thrombosis syndrome.
   9. Current or history of acute polyneuropathy e.g. Guillain-Barré syndrome
   10. Current or history of CDC Category C event
6. Active or chronic hepatitis B virus infection (detectable HBsAg, HBV DNA, or both)
7. Hepatitis C infection (HCV antibody positive)
8. Receipt of a licensed or Emergency Use Authorization vaccine within 4 weeks prior to study screening or plans to receive live attenuated vaccines within 4 weeks or any other licensed or Emergency Use Authorization vaccine within 2 weeks prior to or 2 weeks after any of the study investigational product administrations.
9. Receipt of an investigational study agent within 12 months prior to study screening
10. Previous receipt of immunoglobulin (IgG) therapy Note: Individuals who received IgGs as prophylactic therapy (i.e., for HBV or rabies exposure) >12 months prior to screening will not be excluded.
11. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational Note: Individuals who received monoclonal antibody for the prevention and/or treatment of SARS-CoV-2/COVID-19 >12 months prior to screening will not be excluded.
12. Previous participation in a candidate HIV vaccine study or immune prophylaxis for HIV-1 infection with confirmed receipt of active product or with unknown receipt of active product vs placebo (i.e. remains blinded to what was actually received).
13. History of use of any immunomodulatory medications within 6 months of study entry including systemic corticosteroids (>14 days), immunosuppressants, anti-cancer drugs, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immune modulatory effect Note: Topical or inhaled corticosteroids are not prohibited.
14. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines, vaccine products, neomycin, streptomycin, gentamicin or egg products
15. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment
16. History of chronic urticaria requiring daily treatment or a history of chronic or recurrent eczema and/or atopic dermatitis
17. History of splenectomy
18. EKG abnormality within 90 days prior to or at screening, including but not limited to second or third degree atrioventricular (AV) block, prolongation of the QRS complex over 120 ms (regardless of gender or sex), or clinically important arrhythmia that would interfere with the assessment of myocarditis/pericarditis or QTc interval.
19. QTc interval >440 ms within 90 days prior to or at screening
20. Known family history of Long QT Syndrome in a first-degree relative (i.e., parent, offspring, or sibling).
21. Pregnant, breastfeeding or planning to become pregnant while enrolled in this study
22. Major psychiatric illness and/or substance use during the past 12 months that in the opinion of the investigator would preclude participation

Step 2 (ATI) Inclusion Criteria

Participants enrolled in the study may proceed with Step 2 if the meet all the following inclusion criteria:

1. Receipt at least 3 doses of N-803 and all doses of VRC07-523LS, PGDM1400LS, Ad26.Mos4.HIV with A244d11 gp120/ALFQ and MVA-BN HIV with A244d11 gp120/ALFQ in Step 1.
2. Plasma HIV-1 RNA <50 copies/mL at week 47 visit
3. CD4 T-cell count ≥450 cells/mm3 at week 47 visit

   a. NOTE: The CD4 T-cell count can be repeated once, provided that the repeat is done within 4 weeks prior to Step 2 entry.
4. No CDC Category C event after study entry
5. Documented negative hepatitis B virus (HBV) surface antigen (HBsAg) at week 47 visit
6. Documented negative hepatitis C virus (HCV) antibody (anti-HCV) at week 47 visit
7. For persons of childbearing potential, negative pregnancy test at the week 50 visit
8. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy. One contraceptive method must be from the list of highly effective methods listed in section 7.5.3. The second method of contraception must be from the barrier methods also listed in section 7.5.3.
9. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using pre-exposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
10. Willingness to participate in ATI for up to 36 weeks.
11. Willingness to restart ART according to study guidelines.

Step 2 (ATI) Exclusion Criteria

Enrolled participants who meet any of the following criteria will be excluded from moving to Step 2:

1. Virologic failure (two consecutive HIV-1 RNA >1000 copies/mL) after study entry
2. Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during ATI.
3. Receipt of any non-nucleoside reverse transcriptase inhibitor (NNRTI) within 60 days before Step 2 entry.
4. Receipt of long-acting ART such as long-acting cabotegravir (CAB LA) or long-acting rilpivirine (RPV LA) at any point after Step 1 entry.
5. Failure by the participant to attend three consecutive Step 1 study visits.
6. Pregnancy or breastfeeding.
7. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination in PLWH who initiated ART during AHI. | Through month 31
  Occurrence of ≥ grade 3 AE or SAE that are possibly, probably, or definitely related to the IPs during the study. Adverse events will be graded using "DAIDS TABLE FOR GRADING THE SEVERITY OF ADULT AND PEDIATRIC ADVERSE EVENTS (DAIDS AE SEVERITY GRADING TABLE) V2.1, JULY 2017" (https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf), where grade 1 is mild and grade 4 is potentially life threatening.
To evaluate the treatment combination on time to sustain viral rebound to ≥1000 copies/mL for 4 consecutive weeks AND has not declined by >0.2 log10 | Through month 31
  Time (days) from ATI to sustained viral rebound of ≥1000 copies/mL for 4 consecutive weeks AND has not declined by >0.2 log10 from the previous measurement.

SECONDARY OUTCOMES:
To evaluate the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on time to first documented HIV-1 RNA viral rebound of ≥50 copies/mL following ATI. | Through month 31
  Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥50 copies/mL
To evaluate the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on time to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL following ATI. | Through month 31
  Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL
To evaluate the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on the number of participants with plasma HIV RNA <1000 copies/mL at 12 and 24 weeks of ATI. | Through month 31
  The number of participants with plasma HIV RNA <1000 copies/mL at 12 and 24 weeks of ATI
To evaluate the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on time to ART resumption for an HIV-related (virologic, immunologic, or clinical) reason during Step 2. | Through month 31
  Time (days) from ATI to ART resumption during Step 2
To measure the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on HIV RNA levels while on ART. | Through month 31
  HIV RNA levels using single copy assay while on ART
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on total HIV DNA levels prior to ATI | Through month 31
  Total HIV-1 DNA levels
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on magnitude of T cell responses | Through month 31
  Measured by intracellular cytokine staining (ICS) (Unit: Frequency of cytokine positive T cell in total T cells)
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on breadth of T cell responses | Through month 31
  Measured by Enzyme Linked Immunospot Assay (ELISPOT) (Unit: Spot Forming Units per million cells)
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on effector function of T cell responses | Through month 31
  Measured by percentage of lysis in cytotoxic assay
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on proliferation of T cell responses | Through month 31
  Measured by quantification of 5-6-carboxyfluoresceindiacetate Succimidyl ester (CFSE)-low CD4 and CD8 T cells (Unit: Frequency of CFSE-low T cell in total CD4 or CD8 T cells)
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on HIV specific Binding antibodies to HIV-1 | Through month 31
  Measured by ELISA and expressed as geometric mean endpoint titers
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on HIV specific Antibody Dependent Cellular Cytotoxicity (ADCC): | [Time Frame: Through month 31]
  Measured by ADCC assay expressed as percent lysis of labelled target cells using patient sera versus controls.
To assess the effects of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on HIV specific Antibody Dependent Cellular Phagocytosis (ADCP): | [Time Frame: Through month 31]
  Measured as sample phagocytosis score compared to control.
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on cell-associated HIV DNA prior to ATI | [Time Frame: Through month 31]
  Measured as HIV DNA copies per million PBMC
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on cell-associated HIV RNA prior to ATI | [Time Frame: Through month 31]
  Measured as HIV RNA copies per million PBMC
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on the HIV reservoir prior to ATI using Total Virus Recovery | [Time Frame: Through month 31]
  Measured as HIV nucleic acid copies per million PBMC
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on the HIV reservoir prior to ATI using Intact Proviral DNA: | [Time Frame: Through month 31]
  Measured as the number of intact proviral genomes per million PBMC
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on the HIV reservoir prior to ATI using single copy HIV RNA | [Time Frame: Through month 31]
  Measured as intact proviral DNA copies per million PBMC
To assess the impact of VRC07-523LS, PGDM1400LS and N-803 in combination with Ad26.Mos4.HIV, MVA-BN-HIV and A244d11 gp120/ALFQ vaccination on the HIV reservoir prior to ATI using Quantitative Viral Outgrowth Assay (QVOA) | [Time Frame: Through month 31]
  Measured as Infectious Units Per Million PBMC (IUPM)
To characterize the pharmacokinetics of VRC07-523LS and PGDM1400LS | [Time Frame: Through month 31]
  Levels of VRC07-523LS and PGDM1400LS

CONTACTS AND LOCATIONS:
Overall Officials: Donn Colby, M.D., M.P.H., Study Chair — US Military HIV Research Program; Kiat Ruxrungtham, MD, Principal Investigator — King Chulalongkorn Memorial Hospital
Locations (2):
- Thailand (2):
  - Thai Red Cross AIDS Research Centre (TRCARC), Pathum Wan, Bangkok
  - The Faculty of Medicine, Chulalongkorn University/ King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok

IPD SHARING:
Plan to Share IPD: No